CLINICAL TRIAL: NCT04595162
Title: A Study of GC019F CAR-T Cell Immunotherapy for Relapsed or Refractory B-cell Acute Lymphoblastic Leukemia
Brief Title: A Study of GC019F CAR-T Cell Immunotherapy for Relapsed or Refractory B- ALL
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Gracell Biotechnology Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGC0005
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2019-11

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T treatment group (Experimental): The patients will receive one dose of GC019F.
  Interventions: Biological: GC019F

INTERVENTIONS:
Biological: GC019F — GC019F is the CAR-T cell immunotherapy targeted CD19. The subjects will receive one single infusion of GC019F.

SUMMARY:
The study is an early, open, single-centered trial. The aim of this study is to evaluate the safety and tolerance of GC019F CAR-T cell immunotherapy in relapsed or refractory B-ALL. The study will include 6-12 subjects to receive GC019F therapy.

DETAILED DESCRIPTION:
This study is an early, open, single-centered trial. The major aim of this study is to evaluate the safety and tolerance of GC019F CAR-T cell immunotherapy in relapsed or refractory B-ALL. The study will include 6-12 subjects to receive GC019F single infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years;
2. Eastern cooperative oncology group (ECOG) performance status of 0 to 2;
3. Life expectancy≥12 weeks;
4. CD19 tumor expression demonstrated in bone marrow or peripheral blood by flow cytometry;
5. Relapsed or refractory B- ALL: a) Refractory B- ALL: Fail to achieve a CR after 2 cycles of a standard induction chemotherapy regimen or one-line/multi-line salvage chemotherapy; b) Relapsed B- ALL: Relapse after remission for the first time in 12 months or relapse after one-line/multi-line salvage chemotherapy; Relapse is defined as recurrence of primitive cell in peripheral blood or bone marrow(>5%) after remission; c)Relapse after autologous stem cell transplantation or allogeneic hematopoietic stem cell transplantation; d)Patients with Philadelphia chromosome positive(Ph+) ALL were eligible if they were intolerant to or had failed two lines of tyrosine kinase inhibitor (TKI) therapy, or had t315i mutation.
6. Did not receive hematopoietic stem cell transplantation≤6 months prior to enrollment;
7. Adequate organ function defined as: a) Creatinine clearance (as estimated by Cockcroft Gault method) >60 mL/min; b) Serum ALT/AST <2.5 ULN; c) Total bilirubin <1.5 ULN (subjects with Gilbert's syndrome≤3 ULN); d) Cardiac ejection fraction≥50%, no evidence of clinically significant pericardial effusion as determined by an ECHO; e) No clinically significant pleural effusion; f) Baseline oxygen saturation >92% on room air;
8. Females of reproductive age must be in non-lactation period. Females of childbearing potential must have a negative serum or urine pregnancy test. All subjects must use medical-approved-contraception (such as intrauterine device and contraceptive drugs) during the treatment and in 2 years after cell transfusion treatment; Males should avoid sperm donation;
9. Venous access can be established, peripheral blood mononuclear cells (PBMC) can be collected in researcher's judgement;
10. The subject agrees to and sign informed consent form;
11. The subject can communicate well with the researcher, is willing and able to comply with the research plans, and finish the research according to the research rule.

Exclusion Criteria:

1. Isolated extramedullary leukemia or isolated extramedullary disease relapse;
2. Central nervous system leukemia involved CNS3;
3. Concomitant malignancy other than cured non-melanoma skin cancer or cervical carcinoma in situ or localized prostate cancer or superficial bladder cancer or ductal carcinoma in situ or diagnosis of other malignancy exceeds 5 years without relapse or treatment during the 5 years;
4. Any result of the following infectious disease tests is positive: HIV; HCV; HBsAg; or HBcAb positive with HBV DNA copies positive; TPPA;
5. Live vaccine ≤4 weeks prior to enrollment;
6. For Ph+ ALL, TKI therapy ≤1 week prior to enrollment;
7. History of anti-CD19 therapy or CAR-T or other gene-editing T cell therapy;
8. Presence of ≥ grade 2 acute graft-versus-host disease (GVHD, Glucksberg criteria) or extensive chronic GVHD (Seattle criteria) that require treatment ≤4 weeks prior to enrollment, or during the study period the subject is required to receive anti-GCHD therapy in researcher's judgement;
9. Presence of concomitant disease that require systemic steroids or other immune suppressive therapy during the study period in researcher's judgement; Allogeneic cell therapy (such as donor lymphocyte infusion, DLI) ≤4 weeks prior to enrollment;
10. CNS stereotactic radiotherapy ≤4 weeks prior to enrollment;
11. Toxicities related to previous therapy did not relieved to ≤1 grade, except hematological toxicity and alopecia;
12. Known life-threatening hypersensitivity to cyclophosphamide or fludarabine, or presence of other intolerant conditions, or severe allergic constitution;
13. Patients with active autoimmune disease (e.g., systemic lupus erythematosus, sjogren syndrome, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, Hashimoto's thyroiditis, hypothyroidism which can be controlled by thyroid hormone replacement therapy is an exception);
14. For patients that underwent or plan to undergo major surgical operation before CAR-T treatment, major surgery which required general anesthesia happened ≤4 weeks prior to enrollment, or did not be fully recovered and clinically stable prior to enrollment, or be anticipated to undergo major surgical operation which requires general anesthesia during the study;
15. Took drug from other research≤28 days prior to enrollment;
16. Any unstable cardiovascular diseases happened ≤6 months prior to enrollment, including but not limited to, unstable angina, myocardial infarction, heart failure (NYHA grade≥ III grade), severe arrhythmia that require drug interference, cardiac angioplasty/coronary stent implantation/ cardiac bypass surgery ≤6 months prior to enrollment;
17. Presence of central nervous system (CNS) disease or disease history, including epilepsy, cerebral ischemia/bleeding, dementia, cerebellar disease, or any autoimmune diseases that involve CNS;
18. Any other condition that researcher think it is inappropriate for the subject to anticipate the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2035-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events(AE) | 15 years
  AEs will be collected and graded according to ASTCT consensus(for Cytokine Release Syndrome, CRS and Immune Effector Cell-Associated Neurotoxicity Syndrome, ICANS) and CTCAE v5.0(for AE except for CRS/ICANS )

SECONDARY OUTCOMES:
CAR copies and concentration of GC007F in peripheral blood, bone marrow and CSF | 2 years
  GC007F CAR copies and cells in peripheral blood, bone marrow and CSF will be measured by qPCR and FCM in 2 years
Overall response rate (ORR) and minimal residual disease negative (MRD-) rate of patients who received GC007F infusion | 2 years
  ORR will be estimated as the percentage of patients who achieved CR or CRi. MRD- rate will be estimated as the percentage of patients who achieved MRD-(blast cells in bone marrow<10^-4 as determined by FCM).
Duration of response (DOR), progression-free survival (PFS), overall survival (OS) of patients who received GC007F infusion | 15 years
  DOR refers to the time interval from the date when the patient was evaluated as CR/CRi for the first time to the date when the patient was evaluated as disease relapse or death due to any reason. PFS refers to the time interval from the date of GC007F infusion to the date when the patient was evaluated as disease relapse or death due to any reason. OS refers to the time interval from the date of GC007F infusion to the date when the patient died due to any reason.
Concentration of anti-GC007F antibody after infusion | 2 years
  After GC007F infusion, GC007F antibody in peripheral blood will be measured in 2 years